CLINICAL TRIAL: NCT02608918
Title: An Open-Label Taste Assessment of BMS-955176 in Healthy Subjects
Brief Title: Taste Properties of HIV Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Senopsys, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 206301; AI468-065 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — BMS-955176

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-955176 (Experimental): BMS-955176 specified dose on specified days
  Interventions: Drug: BMS-955176

INTERVENTIONS:
Drug: BMS-955176
  Other Names: HIV Maturation Inhibitor

SUMMARY:
The purpose of the study is to assess the taste properties of HIV inhibitor

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men and women of non-childbearing potential professional sensory panelists
* Aged between 25 and 80 years

Exclusion Criteria:

* History of relevant drug or food allergies, cardiovascular or Central nervous system (CNS) disease, clinically significant pathology, history of mental illness
* Positive HIV test

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
Taste properties of HIV Inhibitor will be measured using the Flavor Profile of the Flavor Leadership Criteria | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Viiv Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Woburn, Massachusetts, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx